CLINICAL TRIAL: NCT05805475
Title: Effects of Tracheal Suctioning With or Without Expiratory Pause Maneuver in Children Submitted to Invasive Mechanical Ventilation: a Randomized Crossover Clinical Trial
Brief Title: Tracheal Suctioning With or Without Expiratory Pause Maneuver in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022-0072
Record Dates: First submitted 2023-03-14; First posted 2023-04-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Mechanical Ventilation Complication; Pediatric Respiratory Diseases
Keywords: Pediatric Critical Care; Respiratory Mechanics; Tracheal Suctioning; Mechanical ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal suctioning without expiratory pause (Active Comparator): Conventional endotracheal suctioning in closed suction system
  Interventions: Other: Endotracheal suctioning without expiratory pause
- Endotracheal suctioning with expiratory pause (Experimental): Endotracheal suctioning in closed suction system associated with expiratory pause maneuver
  Interventions: Other: Endotracheal suctioning with expiratory pause

INTERVENTIONS:
Other: Endotracheal suctioning with expiratory pause — Perform closed endotracheal suctioning with an expiratory pause of 5 seconds
  Arms: Endotracheal suctioning with expiratory pause
Other: Endotracheal suctioning without expiratory pause — Perform closed endotracheal suctioning without expiratory pause
  Arms: Endotracheal suctioning without expiratory pause

SUMMARY:
The purpose of this study is to evaluate the efficacy of tracheal suctioning associate with expiratory pause maneuver in children on invasive mechanical ventilation.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all parents or guardians giving written informed consent will be evaluate for study entry. Children in invasive mechanical ventilation who meet eligibility criteria will be submitted of two techniques of tracheal suctioning (with and without expiratory pause maneuver), randomized in a crossover trial in a 1:1 ratio, for determine the first technique to be applied.

Clinical data will be collected (sex, age, presence of previous disease, diagnosis of hospitalization), as well as the ventilatory parameters (ventilation mode, peak inspiratory pressure, positive end-expiratory pressure, tidal volume, respiratory frequency, fraction of inspired oxygen).

The protocol consists of an initial conventional tracheal suctioning with a negative pressure of 40mmHg for all the participants. After two (2) hours the first technique will be applied and an interval of another two hours for the application of the second technique. Respiratory mechanics and hemodynamic parameters will be evaluate before and after 30 minutes of each tracheal suctioning techniques.

In case of clinical alterations that may aggravate the patients condition during the protocol (oxygen saturation < 85%, heart rate > 190bpm and/or decrease 20% of mean arterial blood pressure), the technique will be interrupted immediately and the patient will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children at invasive mechanical ventilation for more than 24 hours;
* Under the effect of neuromuscular blocker (level of sedation assessed using the Comfort B Scale with a score <10 and without a cough reflex);
* Endotracheal suctioning in a period > 2h before the application of the technique.

Exclusion Criteria:

* Patients with undrained pneumothorax or hemothorax, or presence of subcutaneous emphysema;
* Hemodynamic instability (hypotension refractory to treatment)
* Need of frequent endotracheal suctioning

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Weight of endotracheal suctioning | Immediately after suctioning
  Weight of endotracheal suctioning in milligrams

SECONDARY OUTCOMES:
Peak inspiratory pressure | Baseline and 30 minutes
  Peak inspiratory pressure in centimeters of water (cmH2O)
Plateau pressure | Baseline and 30 minutes
  Plateau pressure in centimeters of water (cmH2O)
Tidal volume | Baseline and 30 minutes
  Tidal volume in milliliters (ml)
Dynamic compliance | Baseline and 30 minutes
  Dynamic compliance in milliliters per kilograms per centimeters of water (mL/kg/cmH2O)
Airway resistance | Baseline and 30 minutes
  Inspiratory and expiratory resistance in centimeters of water per liter (cmH2O/L)
Auto-positive end-expiratory pressure (auto-PEEP) | Baseline and 30 minutes
  Auto-PEEP in centimeters of water (cmH2O)

OTHER OUTCOMES:
Heart rate | Baseline, immediately after suctioning and after 30 minutes
  Heart rate in beats per minute (bpm)
Arterial blood pressure | Baseline, immediately after suctioning and after 30 minutes
  Systolic and diastolic blood pressure in millimeters of mercury (mmHg)
Oxygen saturation | Baseline, immediately after suctioning and after 30 minutes
  Oxygen saturation in percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Ziegler, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No